CLINICAL TRIAL: NCT07389772
Title: INVESTIGATION OF THE EFFECT OF DIFFERENT ACTIVATION TECHNIQUES ON TLR9, IL6, IL10, TNF-ALFA LEVELS IN HEALTHY AND TYPE 2 DIABETIC PATIENTS WITH APICAL PERIODONTITIS REQUIRING RETREATMENT
Acronym: TLR9 in T2DM
Status: Enrolling by invitation | Type: Observational
Sponsor: bengisu yüksel (Other)
Responsible Party: Sponsor-Investigator, bengisu yüksel, phd student, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: 2025.10.03
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healty group: Patients included in the study will be randomly assigned to two main groups using www.randomizer.org.
  DOS samples will be collected in both the control and experimental groups during both sessions. A total of 90 patients will be divided into two main groups: systemically healthy individuals (n=45) and patients with type 2 diabetes (n=45). Each main group will be divided into three subgroups (n=15) according to the irrigation protocol applied: conventional irrigation, ultrasonic activation , and SWEEPS laser activation . Periapical exudate samples will be collected from all patients in both sessions.
- type 2 diabet mellitus group: Patients included in the study will be randomly assigned to two main groups using www.randomizer.org.
  DOS samples will be collected in both the control and experimental groups during both sessions. A total of 90 patients will be divided into two main groups: systemically healthy individuals (n=45) and patients with type 2 diabetes (n=45). Each main group will be divided into three subgroups (n=15) according to the irrigation protocol applied: conventional irrigation, ultrasonic activation , and SWEEPS laser activation . Periapical exudate samples will be collected from all patients in both sessions.

SUMMARY:
The subject of this thesis study is the effects of SWEEPS laser and ultrasonic activation methods on the immune response in the treatment of apical periodontitis in healthy individuals and patients with Type 2 diabetes requiring retreatment, based on a comparative investigation of Toll-like Receptor 9 (TLR-9), Interleukin-6 (IL-6) and Tumour Necrosis Factor alpha (TNF-α), and Interleukin-10 (IL-10) levels.

DETAILED DESCRIPTION:
Patients included in the study will be randomly assigned to two main groups using www.randomizer.org.

DOS samples will be collected in both the control and experimental groups during both sessions. A total of 90 patients will be divided into two main groups: systemically healthy individuals (n=45) and patients with type 2 diabetes (n=45). Each main group will be divided into three subgroups (n=15) according to the irrigation protocol applied: conventional irrigation, ultrasonic activation (16) and SWEEPS laser activation (17) will not be applied, and periapical exudate samples will be taken from all patients in both sessions.

GROUP 1- Healthy patients Group 1A - Conventional irrigation Group 1B - Ultrasonic activation

Group 1C - SWEEPS laser activation

GROUP 2 - Patients with type 2 diabetes Group 2A - Conventional irrigation Group 2B - Ultrasonic activation Group 2C - SWEEPS laser activation

After collecting DOS samples from the relevant teeth, patients will be administered local anaesthesia with 1.8 ml articaine HCl (Ultracain DS Forte; Pharma Vision San. Ve Tic. A.Ş. Istanbul, Turkey) containing 1:100,000 epinephrine, and the teeth will be isolated using a rubber dam. After disinfecting the crowns of the relevant teeth with 2.5% NaOCl, the caries and existing restorations will be removed, and the access cavity will be disinfected with 2.5% NaOCl. After determining the root canal orifices, Protaper Universal Retreatment (Dentsply Mallefer, Ballagues, Switzerland) will be used for root canal filling removal. (18) Subsequently, the working length will be determined using an electronic apex locator (Ai-Pex, Woodpecker Medical Instrument Co., Guilin, China) and confirmed with a periapical radiograph. For the canal shaping procedure, Eighteeth (Changzhou Sifary Medical Technology Co., Ltd., China) endodontic motor and Protaper Gold (Dentsply Sirona, Charlotte, NC, USA) nickel-titanium rotary files, using the crown-down technique, up to #F5.

After each file change, the root canal will be irrigated with 2 mL of 2.5% NaOCl. After the root canal enlargement procedure is completed, the following solutions will be applied for final irrigation: 10 mL of 2.5% NaOCl, 10 mL of 0.5% sodium thiosulphate, 5 mL of distilled water, 5 mL of 17% EDTA, and 5 mL of serum.

After the sample collection process is completed, ELISA analysis will be performed using commercial kits to measure TNF-α, IL-6, IL-10, and TLR-9 levels.

The analysis of the samples will be carried out at the Laboratory of the Scientific and Technological Research Application and Research Centre at Kırıkkale University.

ELISA analysis methods will be performed according to the manufacturer's application instructions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study:

  1. Patients aged 18-50 years
  2. Patients with ASA I status
  3. Patients with Type 2 diabetes whose HbA1c values are between 5.5% and 9.0%, with diabetes diagnosis confirmed by medical history and laboratory tests (HbA1c test)
  4. Upper and lower incisors and lower premolars with chronic apical periodontitis,
  5. Teeth requiring retreatment with a PAI score ≥3 will be included in the study. (15)

Exclusion criteria:

1. ASA II or higher,
2. Pregnant women or those suspected of being pregnant,
3. Patients with localized or generalized periodontitis,
4. Patients with inflammatory or autoimmune diseases such as hepatitis, HIV infection, immunosuppressive chemotherapy, bleeding disorders, Behçet's syndrome, and arthritis,
5. Individuals with HbA1c levels above 9%,

5. Those who have used antibiotics within the last month and anti-inflammatory drugs within the last week, 6. Smokers, 7. Patients with periodontal pockets greater than 3 mm in the relevant tooth, 8. Those with internal or external root resorption, 9. Those with swelling, palpation pain, or a fistula in the relevant area, 10. Those with root fracture or incomplete root formation, 11. Teeth that cannot be isolated with a rubber dam will not be included in the study.

The name, surname, age, gender, contact information, and tooth number to be treated of patients included in the study will be recorded on the case report form. Periapical radiographs will be taken of the relevant teeth prior to root canal treatment to examine the root canal anatomy. The periapical health status of each tooth will be assessed using the PAI score.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include patients aged 18-64 years who present to the Department of Endodontics, Faculty of Dentistry, Kırıkkale University, with an indication for root canal therapy and are diagnosed with either a healthy group(Group 1) or type 2 diabet mellitus (Group 2).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
TLR9 expression levels in periapical exudate and gingival crevicular fluid samples | Immediately after the procedure
  TLR9 will be measured in periapical exudate and gingival crevicular fluid (GCF) samples obtained during routine root canal treatment. The analysis will be performed using the ELISA method. The aim is to compare expression levels between healthy individuals and patients with type 2 diabetes mellitus.

SECONDARY OUTCOMES:
Correlation analysis between TLR9, IL6, IL10, and TNF-α levels in periapical exudate and gingival crevicular fluid samples | Immediately after the procedure
  This study will evaluate the correlation of TLR9, IL6, IL10, and TNF-α within and between two groups, namely healthy individuals and patients diagnosed with type 2 diabetes mellitus, under different irrigation protocols. Using appropriate statistical methods to examine the intra-group and inter-group relationships between biomarkers in pulp tissue, dentin fluid, and gingival crevicular fluid samples, correlation analyses will be performed separately for each group and comparatively between groups.

CONTACTS AND LOCATIONS:
Overall Officials: dilek hancerliogulları, associate professor, Study Director — Kırıkkale University
Locations (1):
- Kirikkale University Faculty of Dentistry, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No